CLINICAL TRIAL: NCT01437215
Title: Prospective, Multicenter, Single Arm Feasibility and Initial Safety Study of the Endologix Fenestrated Stent Graft System for the Endovascular Repair of Juxtarenal/Pararenal (JAA/PAA) Aneurysms
Brief Title: Pilot Study of the Endologix Fenestrated Stent Graft System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0002
Record Dates: First submitted 2011-09-17; First posted 2011-09-20 (Estimated); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Juxtarenal Aortic Aneurysm; Pararenal Aortic Aneurysm
Keywords: aneurysm; renal stent; juxtarenal; pararenal
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fenestrated Endografting (Experimental)
  Interventions: Device: Ventana Fenestrated Stent Graft System

INTERVENTIONS:
Device: Ventana Fenestrated Stent Graft System — Endovascular repair of juxtarenal or pararenal aortic aneurysm

SUMMARY:
The purpose of this study is to determine whether the Endologix fenestrated stent graft system is safe and feasible in the endovascular repair of juxtarenal or pararenal aortic aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent understood and signed and pt agrees to all follow-up visits;
* Abdominal aortic aneurysm with diameter ≥5cm or ≥4cm which has increased by 0.5cm or more in the past six months
* Adequate iliac/femoral access compatible with the required delivery systems
* Non-aneurysmal infrarenal aortic neck <15mm in length
* Most caudal renal artery to aortoiliac bifurcation length at least 70mm
* Proximal non-aneurysmal aortic neck below the SMA with: diameter 18 to 34 mm; length at least 15 mm; angle (clock face) <60° to the aneurysm sac;
* Angle <60° (clock face) between the SMA and celiac artery
* Renal arteries both distal to the SMA by 0-35mm, within 30mm of each other axially, with 4 to 8mm lumen diameter, and with clockface angle of 90° to 210° to each other
* Iliac anatomy suitable for commercial bifurcated stent graft;
* Minimum 3cm overlap achievable between fenestrated and bifurcated stent grafts

Exclusion Criteria:

* Life expectancy <1 year as judged by the investigator;
* Psychiatric or other condition that may interfere with the study;
* Participating in the enrollment or 30-day follow-up phase of another clinical study;
* Known allergy to any device component;
* Coagulopathy or uncontrolled bleeding disorder;
* Contraindication to contrast media or anticoagulants;
* Ruptured, leaking, dissecting, or mycotic aneurysm;
* Serum creatinine (S-Cr) level >2.0 mg/dL;
* Traumatic vascular injury;
* Active systemic or localized groin infection;
* Connective tissue disease (e.g., Marfan's Syndrome);
* Recent (within prior three months) cerebrovascular accident or myocardial infarction;
* Prior renal transplant;
* Length of either renal artery to be stented <13mm;
* Significant occlusive disease or calcification of either renal artery;
* An essential accessory renal artery;
* Indispensable inferior mesenteric artery;
* Untreated aneurysmal disease of the descending thoracic aorta;
* Clinically significant mural thrombus circumferentially in the suprarenal segment;
* Prior iliac artery stent implanted that may interfere with delivery system introduction;
* Unsuitable vascular anatomy
* Pregnancy (female patient of childbearing potential only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-11-02 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Safety - Number of Major Adverse Events (MAEs) | 30 Days
  Major Adverse Events = all cause death; bowel ischemia; myocardial infarction; paraplegia; renal failure; respiratory complications of stroke; blood loss >1000cc
Feasibility- Number of subjects with procedural success (stent graft patency) and absence of type I/III endoleaks or migration | 30 Days
  Procedural Success with aortic/fenestrated and renal stent graft patency and absence of Type I/III endoleak or migration

SECONDARY OUTCOMES:
Safety - Number of Major Adverse Events (MAEs) | >30 Days to 5 Years
  Major Adverse Events = all cause death; bowel ischemia; myocardial infarction; paraplegia; renal failure; respiratory complications of stroke; blood loss >1000cc
Adverse Events | Procedurally to 5 Years
  All adverse events, whether serious or non-serious
Distal Blood Flow | Discharge to 5 Years
  Ankle-brachial index measurements
Renal Dysfunction | Discharge to 5 Years
  eGFR reduction >30% from baseline
Device Performance | 30 Days to 5 Years
  Aortic, fenestrated, and renal stent graft integrity and patency; migration; endoleak; and aneurysm sac morphology

CONTACTS AND LOCATIONS:
Locations (2):
- Pontificia Universidad Católica de Chile, Santiago, Chile
- Auckland City Hospital, Auckland, New Zealand

REFERENCES:
- [Derived] Holden A, Mertens R, Hill A, Marine L, Clair DG. Initial experience with the Ventana fenestrated system for endovascular repair of juxtarenal and pararenal aortic aneurysms. J Vasc Surg. 2013 May;57(5):1235-45. doi: 10.1016/j.jvs.2012.10.125. Epub 2013 Mar 5. PMID 23466185